CLINICAL TRIAL: NCT00652743
Title: Immunogenicity of GSK Biologicals' Pandemic Influenza Vaccine (GSK1562902A) at Different Boosting Vaccination Schedules
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 111443; 111470; 111471; 111472
Record Dates: First submitted 2008-03-21; First posted 2008-04-04 (Estimated); Results first posted 2018-08-02 (Actual); Last update posted 2018-08-02 (Actual); Status verified 2018-06

CONDITIONS: Influenza
Keywords: immunogenicity; safety; GSK pandemic candidate vaccine
MeSH Terms: conditions — Influenza, Human

ARMS (3):
- GSK1562902A M6 Group (Experimental): Healthy male or female adults, primed with 2 doses of adjuvanted investigational H5N1 vaccine (A/Vietnam/1194/04 strain) and boosted 6 months (M6) after primary vaccination with one dose of Pandemic influenza candidate vaccine (GSK1562902A) in study 109630 (NCT00449670), administrated intramuscularly (IM) in the deltoid region of the non-dominant arm.
  Interventions: Biological: Pandemic influenza vaccine GSK1562902A
- GSK1562902A M12 Group (Experimental): Healthy male or female adults, primed with 2 doses of adjuvanted investigational H5N1 vaccine (A/Vietnam/1194/04 strain) in study 109630 (NCT00449670) receiving one dose of Pandemic influenza candidate vaccine (GSK1562902A) in this booster study, at 12 Months (M12) after the primary vaccination, administrated intramuscularly (IM) in the deltoid region of the non-dominant arm.
  Interventions: Biological: Pandemic influenza vaccine GSK1562902A
- GSK1562902A M36 Group (Experimental): Healthy male or female adults, primed with 2 doses of adjuvanted investigational H5N1 vaccine (A/Vietnam/1194/04 strain) in study 109630 (NCT00449670) receiving one dose of Pandemic influenza candidate vaccine (GSK1562902A) in this booster study, at 36 Months (M36) after the primary vaccination, administrated intramuscularly (IM) in the deltoid region of the non-dominant arm.
  Interventions: Biological: Pandemic influenza vaccine GSK1562902A

INTERVENTIONS:
Biological: Pandemic influenza vaccine GSK1562902A — IM administration

SUMMARY:
Today, the leading contender for the next influenza pandemic is H5N1, a strain of avian virus found primarily in domestic and wild birds. Experts warn that the next influenza pandemic is imminent and could be severe. Prevention and control will depend on the rapid production and worldwide distribution of specific pandemic vaccines. Candidate 'pandemic-like' vaccines must be developed and tested in clinical trials to determine the best formulation and vaccination schedule.

The purpose of this study is to assess the immune response of a candidate pandemic vaccine. The protocol posting deals with objectives & outcome measures of the secondary phase of this study. The objectives and outcome measures of the primary phase are presented in a separate protocol posting (NCT number = 00449670).

ELIGIBILITY:
Inclusion Criteria:

* Subjects who completed participation in primary phase of this study.
* Subjects who the investigator believes can and will comply with the requirements of the protocol should be enrolled in the study.
* Written informed consent obtained from the subject.
* Healthy subjects as established by medical history and clinical examination before entering into the study.
* If the subject is female, she must be of non-childbearing potential or be post-menopausal; if of childbearing potential, she must practice adequate contraception for 30 days prior to vaccination, have a negative pregnancy test and continue such precautions for two months after completion of the vaccination series.

Exclusion Criteria:

* Administration of any licensed vaccines within 4 weeks prior to enrolment in this study.
* Planned administration of a vaccine not foreseen by the study protocol: 4 weeks prior to any visit or within 30 days after vaccination.
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within six months prior to the first visit or planned use during the study
* Any confirmed or suspected immunosuppressive or immunodeficient condition, or autoimmune diseases such as Guillain Barre Syndrome, based on medical history and physical examination (no laboratory testing required).
* History of hypersensitivity to vaccines.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine.
* History of chronic alcohol consumption and/or drug abuse.
* Acute clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by physical examination or laboratory screening tests.
* Serious chronic disease including any medically significant chronic pulmonary, cardiovascular, renal, neurological, psychiatric or metabolic disorder, as determined by medical history and physical examination.
* Acute disease at the time of enrolment.
* Administration of immunoglobulins and/or any blood products within the three months preceding the first visit or planned use during the study.
* Pregnant or lactating women.
* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine(s) within 30 days prior to the first visit, or planned use during the study period.
* Any condition which, in the opinion of the investigator, prevents the subject from participation in the study.

Ages: 19 Years to 61 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 845 (Actual)
Dates: Start 2008-03-23 (Actual); Primary Completion 2011-06-08 (Actual); Study Completion 2011-06-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (4):
- GSK Investigational Site, Hong Kong, Hong Kong
- GSK Investigational Site, Singapore, Singapore
- GSK Investigational Site, Taipei, Taiwan
- GSK Investigational Site, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Gillard P, Chu DW, Hwang SJ, Yang PC, Thongcharoen P, Lim FS, Drame M, Walravens K, Roman F. Long-term booster schedules with AS03A-adjuvanted heterologous H5N1 vaccines induces rapid and broad immune responses in Asian adults. BMC Infect Dis. 2014 Mar 15;14:142. doi: 10.1186/1471-2334-14-142. PMID 24628789
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 111443 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 111443 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register. The results of this study 111470 are summarised with studies 111443, 111471, and 111472 on the GSK Clinical Study Register.
- Available data/document: Study Protocol: 111443 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 111443 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 111443 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 111443 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One enrolled subject was not administered a booster vaccination and hence not considered to have started the study.
Period: Months 12-18
Arm/Group | GSK1562902A M6 Group | GSK1562902A M12 Group | GSK1562902A M36 Group
Started | 219 | 188 | 437
Completed | 218 | 186 | 430
Not Completed | 1 | 2 | 7
Not completed — Lost to Follow-up | 1 | 2 | 7
Period: Months 24-30
Arm/Group | GSK1562902A M6 Group | GSK1562902A M12 Group | GSK1562902A M36 Group
Started | 212 | 186 | 433
Completed | 207 | 185 | 422
Not Completed | 5 | 1 | 11
Not completed — Other | 5 | 1 | 11
Period: Months 36-42
Arm/Group | GSK1562902A M6 Group | GSK1562902A M12 Group | GSK1562902A M36 Group
Started | 216 | 185 | 390
Completed | 210 | 180 | 381
Not Completed | 6 | 5 | 9
Not completed — Serious Adverse Events | 0 | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Migrated/moved from study area | 1 | 0 | 0
Not completed — Other | 4 | 2 | 8
Period: Months 42-48
Arm/Group | GSK1562902A M6 Group | GSK1562902A M12 Group | GSK1562902A M36 Group
Started | 196 | 170 | 367
Completed | 196 | 170 | 367
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GSK1562902A M6 Group | GSK1562902A M12 Group | GSK1562902A M36 Group | Total
Number analyzed (Participants) | 219 | 188 | 437 | 844
Age, Continuous [Mean (Standard Deviation); unit: Years] | 34.1 (10.33) | 35.3 (9.23) | 35.4 (9.71) | 34.93 (9.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 113 | 97 | 210 | 420
  Male | 106 | 91 | 227 | 424
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Boosted at Month 12 With Haemagglutinin-inhibition (HI) Antibody Concentrations Above the Cut-off Value
Description: Seropositivity cut-off values assessed were equal to or above (≥) 1:10 in the sera of subjects seronegative before vaccination. The flu strain assessed was Flu A/Indonesia/05/2005.
Time Frame: At Month 12 + 21 days
Population: The analysis was performed on the According-to-Protocol (ATP) cohort for immunogenicity, which included all evaluable subjects for whom immunogenicity data were available. This included subjects for whom assay results were available for antibodies against at least one study vaccine antigen component after vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A M12 Group
Number analyzed (Participants) | 186
Participants | 178

2. Primary Outcome: Titers for Antibodies Against A/Indonesia/05/2005 Strain of Influenza Disease for Subjects Boosted at Month 12
Description: Titers are presented as geometric mean titers (GMTs). The reference seropositivity cut-off value was equal to or above (≥) 1:10. The flu strain assessed was Flu A/Indonesia/05/2005.
Time Frame: At Month 12 + 21 days
Population: The analysis was performed on the ATP cohort for immunogenicity, which included all evaluable subjects for whom immunogenicity data were available. This included subjects for whom assay results were available for antibodies against at least one study vaccine antigen component after vaccination.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | GSK1562902A M12 Group
Number analyzed (Participants) | 186
Titers | 340.3 [282.8 to 409.6]

3. Primary Outcome: Number of Subjects Boosted at Month 36 With HI Antibody Concentrations Above the Cut-off Value
Description: as for outcome 1
Time Frame: At Month 36 + 21 days
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A M36 Group
Number analyzed (Participants) | 379
Participants | 379

4. Primary Outcome: Titers for Antibodies Against A/Indonesia/05/2005 Strain of Influenza Disease for Subjects Boosted at Month 36
Description: as for outcome 2
Time Frame: At Month 36 + 21 days
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | GSK1562902A M36 Group
Number analyzed (Participants) | 379
Titers | 877.5 [809.1 to 951.6]

5. Primary Outcome: Booster Vaccine Response for HI Antibodies Against A/Indonesia/05/2005 Strain of Influenza Disease for Subjects Boosted at Month 12
Description: Booster vaccine response was defined as: antibody titer after booster vaccination ≥ 4-fold the pre-booster antibody titer. The Flu strain assessed was A/Indonesia/05/2005 (H5N1).
Time Frame: At Month 12 + 21 days
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A M12 Group
Number analyzed (Participants) | 180
Participants | 169

6. Primary Outcome: Booster Vaccine Response for HI Antibodies Against A/Indonesia/05/2005 Strain of Influenza Disease for Subjects Boosted at Month 36
Description: as for outcome 5
Time Frame: At Month 36 + 21 Days
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A M36 Group
Number analyzed (Participants) | 379
Participants | 378

7. Primary Outcome: Geometric Mean Fold Rise (GMFR) for HI Antibodies Against A/Indonesia/05/2005 Strain of Influenza Disease for Subjects Boosted at Month 12
Description: GMFR, also known as seroconversion factor (SCF), was defined as the geometric mean of the within-subject ratios of the post-vaccination reciprocal HI titer to the pre-vaccination reciprocal HI titer for the vaccine virus. The flu strain assessed was Flu A/Indonesia/05/2005.
Time Frame: At Month 12 + 21 days
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Fold change
Arm/Group | GSK1562902A M12 Group
Number analyzed (Participants) | 180
Fold change | 55.3 [45.2 to 67.6]

8. Primary Outcome: Geometric Mean Fold Rise (GMFR) for HI Antibodies Against A/Indonesia/05/2005 Strain of Influenza Disease for Subjects Boosted at Month 36
Description: as for outcome 7
Time Frame: At Month 36 +21 days
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Fold change
Arm/Group | GSK1562902A M36 Group
Number analyzed (Participants) | 379
Fold change | 123.8 [112.1 to 136.8]

9. Primary Outcome: Number of Subjects Boosted at Month 12 Seroprotected (SPR) for HI Antibodies Against A/Indonesia/05/2005 Strain of Influenza Disease
Description: Seroprotection (SPR) was defined as the proportion of subjects with H5N1 reciprocal HI titers equal to or above (≥) 1:40 against the tested vaccine virus. The flu strain assessed was Flu A/Indonesia/05/2005.
Time Frame: At Month 12 + 21 days
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A M12 Group
Number analyzed (Participants) | 186
Participants | 178

10. Primary Outcome: Number of Subjects Boosted at Month 36 Seroprotected (SPR) for HI Antibodies Against A/Indonesia/05/2005 Strain of Influenza Disease
Description: as for outcome 9
Time Frame: At Month 36 + 21 days
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A M36 Group
Number analyzed (Participants) | 379
Participants | 379

11. Secondary Outcome: Number of Seropositive Subjects for H5N1 HI Antibodies
Description: Seropositivity was defined as the proportion of subjects with H5N1 reciprocal HI titers equal to or above (≥) 1:10 against the tested vaccine virus. The flu strains assessed were A/Indonesia/05/2005 and A/Vietnam/1194/2004.
Time Frame: At Months 18, 24, 30 and 36
Population: The analysis was performed on the ATP cohort for persistence at Month 12-18 (M12-18) and at Month 24-30 (M24-30), which included all evaluable subjects not boosted (M12-18) and boosted (M24-30) at M12, not boosted at M12 but boosted at M6 or neither boosted at M6 nor at M12 (M24-30).
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A M6 Group | GSK1562902A M12 Group | GSK1562902A M36 Group
Number analyzed (Participants) | 216 | 178 | 429
Participants
  A/Indonesia/05/2005, Month 18: number analyzed (Participants) | 216 | 0 | 429
  A/Indonesia/05/2005, Month 18 | 178 | 0 | 146
  A/Indonesia/05/2005, Month 24: number analyzed (Participants) | 200 | 177 | 411
  A/Indonesia/05/2005, Month 24 | 142 | 147 | 58
  A/Indonesia/05/2005, Month 30: number analyzed (Participants) | 200 | 177 | 413
  A/Indonesia/05/2005, Month 30 | 144 | 149 | 73
  A/Indonesia/05/2005, Month 36: number analyzed (Participants) | 208 | 178 | 0
  A/Indonesia/05/2005, Month 36 | 144 | 147 | 0
  A/Vietnam/1194/2004, Month 18: number analyzed (Participants) | 216 | 0 | 429
  A/Vietnam/1194/2004, Month 18 | 176 | 0 | 173
  A/Vietnam/1194/2004, Month 24: number analyzed (Participants) | 200 | 177 | 411
  A/Vietnam/1194/2004, Month 24 | 161 | 154 | 187
  A/Vietnam/1194/2004, Month 30: number analyzed (Participants) | 200 | 177 | 413
  A/Vietnam/1194/2004, Month 30 | 154 | 158 | 168
  A/Vietnam/1194/2004, Month 36: number analyzed (Participants) | 208 | 178 | 0
  A/Vietnam/1194/2004, Month 36 | 149 | 152 | 0

12. Secondary Outcome: Number of Seropositive Subjects for H5N1 HI Antibodies
Description: as for outcome 11
Time Frame: At Months 42 and 48
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A M6 Group | GSK1562902A M12 Group | GSK1562902A M36 Group
Number analyzed (Participants) | 201 | 176 | 367
Participants
  A/Indonesia/05/2005, Month 42: number analyzed (Participants) | 201 | 176 | 0
  A/Indonesia/05/2005, Month 42 | 127 | 143 | 0
  A/Indonesia/05/2005, Month 48: number analyzed (Participants) | 194 | 170 | 367
  A/Indonesia/05/2005, Month 48 | 125 | 133 | 365
  A/Vietnam/1194/2004, Month 42: number analyzed (Participants) | 201 | 176 | 0
  A/Vietnam/1194/2004, Month 42 | 138 | 149 | 0
  A/Vietnam/1194/2004, Month 48: number analyzed (Participants) | 194 | 170 | 367
  A/Vietnam/1194/2004, Month 48 | 137 | 142 | 365

13. Secondary Outcome: Booster Vaccine Response for H5N1 HI Antibodies for Subjects Boosted at Month 6 and Month 12
Description: Booster vaccine response was defined as: antibody titer after booster vaccination ≥ 4 fold the pre-booster antibody titer. The Flu strains assessed were A/Indonesia/05/2005 and A/Vietnam/1194/2004.
Time Frame: At Months 18, 24 and 30
Population: The analysis was performed on the ATP cohort for persistence at Month 12-18 and at Month 24-30, which included all evaluable subjects not boosted and boosted at Month 12, not boosted at Month 12 but boosted at Month 6 or neither boosted at Month 6 nor at Month 12.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A M6 Group | GSK1562902A M12 Group
Number analyzed (Participants) | 216 | 113
Participants
  A/Indonesia/05/2005, Month 18: number analyzed (Participants) | 216 | 0
  A/Indonesia/05/2005, Month 18 | 149 | 0
  A/Indonesia/05/2005, Month 24: number analyzed (Participants) | 146 | 113
  A/Indonesia/05/2005, Month 24 | 48 | 70
  A/Indonesia/05/2005, Month 30: number analyzed (Participants) | 146 | 113
  A/Indonesia/05/2005, Month 30 | 52 | 69
  A/Vietnam/1194/2004, Month 18: number analyzed (Participants) | 216 | 0
  A/Vietnam/1194/2004, Month 18 | 68 | 0
  A/Vietnam/1194/2004, Month 24: number analyzed (Participants) | 146 | 113
  A/Vietnam/1194/2004, Month 24 | 32 | 61
  A/Vietnam/1194/2004, Month 30: number analyzed (Participants) | 146 | 113
  A/Vietnam/1194/2004, Month 30 | 28 | 51

14. Secondary Outcome: Number of Subjects Boosted at Month 36 Seroconverted for H5N1 HI Antibodies
Description: Seroconversion was defined as the proportion of subjects who had either a pre-vaccination reciprocal HI titer < 10 and a post-vaccination reciprocal titer ≥ 40, or a pre-vaccination reciprocal HI titer ≥ 10 and at least a 4-fold increase in post-vaccination reciprocal titer against the vaccine virus. The flu strains assessed were A/Indonesia/05/2005 and A/Vietnam/1194/2004.
Time Frame: At Months 18, 24 and 30
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A M36 Group
Number analyzed (Participants) | 428
Participants
  A/Indonesia/05/2005, Month 18 | 75
  A/Indonesia/05/2005, Month 24: number analyzed (Participants) | 284
  A/Indonesia/05/2005, Month 24 | 6
  A/Indonesia/05/2005, Month 30: number analyzed (Participants) | 284
  A/Indonesia/05/2005, Month 30 | 14
  A/Vietnam/1194/2004, Month 18 | 61
  A/Vietnam/1194/2004, Month 24: number analyzed (Participants) | 284
  A/Vietnam/1194/2004, Month 24 | 43
  A/Vietnam/1194/2004, Month 30: number analyzed (Participants) | 284
  A/Vietnam/1194/2004, Month 30 | 58

15. Secondary Outcome: Booster Vaccine Response for H5N1 HI Antibodies
Description: Booster vaccine response was defined as: antibody titer after booster vaccination ≥ 4-fold the pre-booster antibody titer. The Flu strains assessed were A/Indonesia/05/2005 and A/Vietnam/1194/2004.
Time Frame: At Months 36, 42 and 48
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A M6 Group | GSK1562902A M12 Group | GSK1562902A M36 Group
Number analyzed (Participants) | 208 | 172 | 367
Participants
  A/Indonesia/05/2005, Month 36: number analyzed (Participants) | 208 | 172 | 0
  A/Indonesia/05/2005, Month 36 | 91 | 115 | 0
  A/Indonesia/05/2005, Month 42: number analyzed (Participants) | 201 | 170 | 0
  A/Indonesia/05/2005, Month 42 | 59 | 89 | 0
  A/Indonesia/05/2005, Month 48: number analyzed (Participants) | 194 | 164 | 367
  A/Indonesia/05/2005, Month 48 | 62 | 88 | 339
  A/Vietnam/1194/2004, Month 36: number analyzed (Participants) | 208 | 172 | 0
  A/Vietnam/1194/2004, Month 36 | 28 | 82 | 0
  A/Vietnam/1194/2004, Month 42: number analyzed (Participants) | 201 | 170 | 0
  A/Vietnam/1194/2004, Month 42 | 22 | 69 | 0
  A/Vietnam/1194/2004, Month 48: number analyzed (Participants) | 194 | 164 | 367
  A/Vietnam/1194/2004, Month 48 | 28 | 75 | 319

16. Secondary Outcome: Geometric Mean Fold Rise (GMFR) for H5N1 HI Antibodies
Description: GMFR, also known as seroconversion factor (SCF), was defined as the geometric mean of the within-subject ratios of the post-vaccination reciprocal HI titer to the pre-vaccination reciprocal HI titer for the vaccine virus. The flu strains assessed were A/Indonesia/05/2005 and A/Vietnam/1194/2004.
Time Frame: At Months 18, 24, 30
Population: as for outcome 13
Measure: Geometric Mean (95% Confidence Interval); unit: Fold change
Arm/Group | GSK1562902A M6 Group | GSK1562902A M12 Group | GSK1562902A M36 Group
Number analyzed (Participants) | 216 | 170 | 428
Fold change
  A/Indonesia/05/2005, Month 18: number analyzed (Participants) | 216 | 0 | 428
  A/Indonesia/05/2005, Month 18 | 8.4 [7.0 to 10.1] |  | 1.9 [1.7 to 2.1]
  A/Indonesia/05/2005, Month 24: number analyzed (Participants) | 200 | 170 | 410
  A/Indonesia/05/2005, Month 24 | 3.4 [2.9 to 4.1] | 8.5 [6.8 to 10.6] | 1.2 [1.1 to 1.2]
  A/Indonesia/05/2005, Month 30: number analyzed (Participants) | 200 | 170 | 412
  A/Indonesia/05/2005, Month 30 | 3.4 [2.9 to 4.0] | 7.6 [6.2 to 9.4] | 1.2 [1.2 to 1.3]
  A/Vietnam/1194/2004, Month 18: number analyzed (Participants) | 216 | 0 | 428
  A/Vietnam/1194/2004, Month 18 | 2.4 [2.0 to 2.9] |  | 1.8 [1.7 to 2.0]
  A/Vietnam/1194/2004, Month 24: number analyzed (Participants) | 200 | 170 | 410
  A/Vietnam/1194/2004, Month 24 | 1.7 [1.5 to 2.1] | 6.1 [4.9 to 7.5] | 1.9 [1.8 to 2.1]
  A/Vietnam/1194/2004, Month 30: number analyzed (Participants) | 200 | 170 | 412
  A/Vietnam/1194/2004, Month 30 | 1.5 [1.3 to 1.8] | 4.8 [4.0 to 5.8] | 1.9 [1.7 to 2.1]

17. Secondary Outcome: Geometric Mean Fold Rise (GMFR) for H5N1 HI Antibodies
Description: as for outcome 16
Time Frame: At Months 36, 42 and 48
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Fold change
Arm/Group | GSK1562902A M6 Group | GSK1562902A M12 Group | GSK1562902A M36 Group
Number analyzed (Participants) | 208 | 172 | 367
Fold change
  A/Indonesia/05/2005, Month 36: number analyzed (Participants) | 208 | 172 | 0
  A/Indonesia/05/2005, Month 36 | 3.8 [3.2 to 4.5] | 8.6 [6.9 to 10.7] |
  A/Indonesia/05/2005, Month 42: number analyzed (Participants) | 201 | 170 | 0
  A/Indonesia/05/2005, Month 42 | 2.8 [2.4 to 3.2] | 6.0 [4.9 to 7.4] |
  A/Indonesia/05/2005, Month 48: number analyzed (Participants) | 194 | 164 | 367
  A/Indonesia/05/2005, Month 48 | 3.0 [2.6 to 3.6] | 6.1 [5.0 to 7.5] | 24.0 [21.5 to 26.9]
  A/Vietnam/1194/2004, Month 36: number analyzed (Participants) | 208 | 172 | 0
  A/Vietnam/1194/2004, Month 36 | 1.3 [1.1 to 1.6] | 4.5 [3.7 to 5.5] |
  A/Vietnam/1194/2004, Month 42: number analyzed (Participants) | 201 | 170 | 0
  A/Vietnam/1194/2004, Month 42 | 1.1 [0.9 to 1.3] | 3.4 [2.8 to 4.1] |
  A/Vietnam/1194/2004, Month 48: number analyzed (Participants) | 194 | 164 | 367
  A/Vietnam/1194/2004, Month 48 | 1.2 [1.0 to 1.5] | 3.7 [3.0 to 4.5] | 15.2 [13.4 to 17.1]

18. Secondary Outcome: Number of Seroprotected (SPR) Subjects for H5N1 HI Antibodies
Description: Seroprotection (SPR) was defined as the proportion of subjects with H5N1 reciprocal HI titers equal to or above (≥) 1:40 against the tested vaccine virus. The flu strains assessed were A/Indonesia/05/2005 and A/Vietnam/1194/2004.
Time Frame: At Months 18, 24 and 30
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A M6 Group | GSK1562902A M12 Group | GSK1562902A M36 Group
Number analyzed (Participants) | 216 | 177 | 429
Participants
  A/Indonesia/05/2005, Month 18: number analyzed (Participants) | 216 | 0 | 429
  A/Indonesia/05/2005, Month 18 | 157 | 0 | 75
  A/Indonesia/05/2005, Month 24: number analyzed (Participants) | 200 | 177 | 411
  A/Indonesia/05/2005, Month 24 | 88 | 117 | 10
  A/Indonesia/05/2005, Month 30: number analyzed (Participants) | 200 | 177 | 413
  A/Indonesia/05/2005, Month 30 | 95 | 120 | 16
  A/Vietnam/1194/2004, Month 18: number analyzed (Participants) | 216 | 0 | 429
  A/Vietnam/1194/2004, Month 18 | 149 | 0 | 79
  A/Vietnam/1194/2004, Month 24: number analyzed (Participants) | 200 | 177 | 411
  A/Vietnam/1194/2004, Month 24 | 115 | 135 | 67
  A/Vietnam/1194/2004, Month 30: number analyzed (Participants) | 200 | 177 | 413
  A/Vietnam/1194/2004, Month 30 | 107 | 128 | 88

19. Secondary Outcome: Number of Seroprotected (SPR) Subjects for H5N1 HI Antibodies
Description: as for outcome 18
Time Frame: At Months 36, 42 and 48
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A M6 Group | GSK1562902A M12 Group | GSK1562902A M36 Group
Number analyzed (Participants) | 208 | 178 | 367
Participants
  A/Indonesia/05/2005, Month 36: number analyzed (Participants) | 208 | 178 | 0
  A/Indonesia/05/2005, Month 36 | 104 | 126 | 0
  A/Indonesia/05/2005, Month 42: number analyzed (Participants) | 201 | 176 | 0
  A/Indonesia/05/2005, Month 42 | 70 | 101 | 0
  A/Indonesia/05/2005, Month 48: number analyzed (Participants) | 194 | 170 | 367
  A/Indonesia/05/2005, Month 48 | 76 | 104 | 351
  A/Vietnam/1194/2004, Month 36: number analyzed (Participants) | 208 | 178 | 0
  A/Vietnam/1194/2004, Month 36 | 90 | 121 | 0
  A/Vietnam/1194/2004, Month 42: number analyzed (Participants) | 201 | 176 | 0
  A/Vietnam/1194/2004, Month 42 | 79 | 110 | 0
  A/Vietnam/1194/2004, Month 48: number analyzed (Participants) | 194 | 170 | 367
  A/Vietnam/1194/2004, Month 48 | 88 | 114 | 349

20. Secondary Outcome: Titers for Serum Neutralizing Antibodies
Description: Titers were presented as geometric mean titers (GMTs). The reference seropositivity cut-off value was equal to or above (≥) 1:28. The flu strains assessed were A/Indonesia/05/2005 and A/Vietnam/1194/2004.
Time Frame: At Months 6/12, 6/12 + 21 days, 24, 36 and 48
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | GSK1562902A M6 Group | GSK1562902A M12 Group | GSK1562902A M36 Group
Number analyzed (Participants) | 163 | 170 | 75
Titers
  A/Indonesia/05/2005, Month 6: number analyzed (Participants) | 162 | 0 | 0
  A/Indonesia/05/2005, Month 6 | 179.7 [161.8 to 199.7] |  |
  A/Indonesia/05/2005, Month 6/12/36 + 21 days: number analyzed (Participants) | 162 | 170 | 75
  A/Indonesia/05/2005, Month 6/12/36 + 21 days | 2702.0 [2270.4 to 3215.6] | 2363.2 [2037.5 to 2740.9] | 1154.3 [847.8 to 1571.4]
  A/Indonesia/05/2005, Month 12: number analyzed (Participants) | 74 | 164 | 0
  A/Indonesia/05/2005, Month 12 | 134.0 [107.4 to 167.3] | 58.5 [50.8 to 67.3] |
  A/Indonesia/05/2005, Month 24: number analyzed (Participants) | 74 | 75 | 75
  A/Indonesia/05/2005, Month 24 | 66.3 [54.5 to 80.8] | 148.9 [111.8 to 198.3] | 16.7 [15.4 to 18.1]
  A/Indonesia/05/2005, Month 36: number analyzed (Participants) | 75 | 74 | 75
  A/Indonesia/05/2005, Month 36 | 55.4 [45.5 to 67.6] | 106.9 [81.6 to 140.0] | 17.3 [15.8 to 19.0]
  A/Indonesia/05/2005, Month 48: number analyzed (Participants) | 75 | 75 | 75
  A/Indonesia/05/2005, Month 48 | 54.5 [45.8 to 64.7] | 103.4 [79.5 to 134.4] | 320.4 [243.7 to 421.4]
  A/Vietnam/1194/2004, Month 6: number analyzed (Participants) | 163 | 0 | 0
  A/Vietnam/1194/2004, Month 6 | 169.9 [152.3 to 189.4] |  |
  A/Vietnam/1194/2004, Month 6/12/36 + 21 days: number analyzed (Participants) | 163 | 170 | 74
  A/Vietnam/1194/2004, Month 6/12/36 + 21 days | 1566.3 [1342.1 to 1827.9] | 2734.9 [2334.4 to 3204.2] | 1373.4 [1023.7 to 1842.6]
  A/Vietnam/1194/2004, Month 12: number analyzed (Participants) | 75 | 164 | 0
  A/Vietnam/1194/2004, Month 12 | 159.4 [128.1 to 198.2] | 204.1 [179.9 to 231.6] |
  A/Vietnam/1194/2004, Month 24: number analyzed (Participants) | 75 | 75 | 75
  A/Vietnam/1194/2004, Month 24 | 74.0 [62.5 to 87.5] | 164.9 [125.7 to 216.2] | 33.3 [28.8 to 38.4]
  A/Vietnam/1194/2004, Month 36: number analyzed (Participants) | 75 | 74 | 75
  A/Vietnam/1194/2004, Month 36 | 62.0 [52.1 to 73.7] | 121.1 [91.7 to 159.9] | 31.8 [27.3 to 36.9]
  A/Vietnam/1194/2004, Month 48: number analyzed (Participants) | 75 | 75 | 75
  A/Vietnam/1194/2004, Month 48 | 71.4 [61.8 to 82.5] | 117.4 [92.7 to 148.6] | 429.0 [322.2 to 571.2]

21. Secondary Outcome: Booster Vaccine Response for Neutralizing Antibodies
Description: Booster vaccine response was defined as: for pre-booster antibody titer < 1:28, antibody titer ≥ 1:56 post-booster; for pre-booster, antibody titer ≥ 1:28, post-booster ≥ 4-fold the pre-booster antibody titer. The flu strains assessed were A/Indonesia/05/2005 and A/Vietnam/1194/2004.
Time Frame: At Months 6/12/36 + 21 days, 12, 24, 36 and 48
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A M6 Group | GSK1562902A M12 Group | GSK1562902A M36 Group
Number analyzed (Participants) | 163 | 164 | 75
Participants
  A/Indonesia/05/2005, Month 12: number analyzed (Participants) | 74 | 0 | 0
  A/Indonesia/05/2005, Month 12 | 4 | 0 | 0
  A/Indonesia/05/2005, Month 24: number analyzed (Participants) | 74 | 75 | 0
  A/Indonesia/05/2005, Month 24 | 0 | 34 | 0
  A/Indonesia/05/2005, Month 36: number analyzed (Participants) | 75 | 74 | 0
  A/Indonesia/05/2005, Month 36 | 0 | 27 | 0
  A/Indonesia/05/2005, Month 48: number analyzed (Participants) | 75 | 75 | 75
  A/Indonesia/05/2005, Month 48 | 1 | 27 | 72
  A/Indonesia/05/2005, Month 6/12/36 + 21 days: number analyzed (Participants) | 162 | 164 | 75
  A/Indonesia/05/2005, Month 6/12/36 + 21 days | 144 | 159 | 75
  A/Vietnam/1194/2004, Month 12: number analyzed (Participants) | 75 | 0 | 0
  A/Vietnam/1194/2004, Month 12 | 7 | 0 | 0
  A/Vietnam/1194/2004, Month 24: number analyzed (Participants) | 75 | 75 | 0
  A/Vietnam/1194/2004, Month 24 | 1 | 7 | 0
  A/Vietnam/1194/2004, Month 36: number analyzed (Participants) | 75 | 74 | 0
  A/Vietnam/1194/2004, Month 36 | 0 | 5 | 0
  A/Vietnam/1194/2004, Month 48: number analyzed (Participants) | 75 | 75 | 75
  A/Vietnam/1194/2004, Month 48 | 0 | 2 | 64
  A/Vietnam/1194/2004, Month 6/12/36 + 21 days: number analyzed (Participants) | 163 | 164 | 74
  A/Vietnam/1194/2004, Month 6/12/36 + 21 days | 121 | 141 | 73

22. Secondary Outcome: Number of Subjects With Neutralizing Antibody Concentrations Above the Cut-off Value
Description: Seropositivity cut-off values assessed were equal to or above (≥) 1:28, ≥ 1:56 and ≥ 1:112 in the sera of subjects seronegative before vaccination. The flu strain assessed was A/Indonesia/05/2005.
Time Frame: At Months 6/12/36 + 21 days, 12, 24, 36 and 48
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A M6 Group | GSK1562902A M12 Group | GSK1562902A M36 Group
Number analyzed (Participants) | 162 | 170 | 75
Participants
  Month 6, ≥ 1:28: number analyzed (Participants) | 162 | 0 | 0
  Month 6, ≥ 1:28 | 160 | 0 | 0
  Month 12, ≥ 1:28: number analyzed (Participants) | 74 | 164 | 0
  Month 12, ≥ 1:28 | 74 | 135 | 0
  Month 24, ≥ 1:28: number analyzed (Participants) | 74 | 75 | 75
  Month 24, ≥ 1:28 | 70 | 72 | 17
  Month 36, ≥ 1:28: number analyzed (Participants) | 75 | 74 | 75
  Month 36, ≥ 1:28 | 66 | 69 | 19
  Month 48, ≥ 1:28: number analyzed (Participants) | 75 | 75 | 75
  Month 48, ≥ 1:28 | 67 | 73 | 74
  Month 6/12/36 + 21 days, ≥ 1:28 | 162 | 170 | 75
  Month 6, ≥ 1:56: number analyzed (Participants) | 162 | 0 | 0
  Month 6, ≥ 1:56 | 153 | 0 | 0
  Month 12, ≥ 1:56: number analyzed (Participants) | 74 | 164 | 0
  Month 12, ≥ 1:56 | 70 | 99 | 0
  Month 24, ≥ 1:56: number analyzed (Participants) | 74 | 75 | 75
  Month 24, ≥ 1:56 | 54 | 67 | 2
  Month 36, ≥ 1:56: number analyzed (Participants) | 75 | 74 | 75
  Month 36, ≥ 1:56 | 48 | 58 | 4
  Month 48, ≥ 1:56: number analyzed (Participants) | 75 | 75 | 75
  Month 48, ≥ 1:56 | 51 | 58 | 72
  Month 6/12/36 + 21 days, ≥ 1:56 | 162 | 170 | 74
  Month 6, ≥ 1:112: number analyzed (Participants) | 162 | 0 | 0
  Month 6, ≥ 1:112 | 140 | 0 | 0
  Month 12, ≥ 1:112: number analyzed (Participants) | 74 | 164 | 0
  Month 12, ≥ 1:112 | 50 | 45 | 0
  Month 24, ≥ 1:112: number analyzed (Participants) | 74 | 75 | 75
  Month 24, ≥ 1:112 | 26 | 47 | 0
  Month 36, ≥ 1:112: number analyzed (Participants) | 75 | 74 | 75
  Month 36, ≥ 1:112 | 24 | 41 | 0
  Month 48, ≥ 1:112: number analyzed (Participants) | 75 | 75 | 75
  Month 48, ≥ 1:112 | 23 | 39 | 65
  Month 6/12/36 + 21 days, ≥ 1:112 | 161 | 170 | 71

23. Secondary Outcome: Number of Subjects With Neutralizing Antibody Concentrations Above the Cut-off
Description: Seropositivity cut-off values assessed were equal to or above (≥) 1:28, ≥ 1:56 and ≥ 1:112 in the sera of subjects seronegative before vaccination. The flu strain assessed was A/Vietnam/1194/2004.
Time Frame: At Months 6/12/36 + 21 days, 12, 24, 36 and 48
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A M6 Group | GSK1562902A M12 Group | GSK1562902A M36 Group
Number analyzed (Participants) | 163 | 170 | 75
Participants
  Month 6, ≥ 1:28: number analyzed (Participants) | 163 | 0 | 0
  Month 6, ≥ 1:28 | 162 | 0 | 0
  Month 12, ≥ 1:28: number analyzed (Participants) | 75 | 164 | 0
  Month 12, ≥ 1:28 | 75 | 162 | 0
  Month 24, ≥ 1:28: number analyzed (Participants) | 75 | 75 | 75
  Month 24, ≥ 1:28 | 74 | 75 | 58
  Month 36, ≥ 1:28: number analyzed (Participants) | 75 | 74 | 75
  Month 36, ≥ 1:28 | 71 | 73 | 55
  Month 48, ≥ 1:28: number analyzed (Participants) | 75 | 75 | 75
  Month 48, ≥ 1:28 | 73 | 74 | 74
  Month 6/12/36 + 21 days, ≥ 1:28: number analyzed (Participants) | 163 | 170 | 74
  Month 6/12/36 + 21 days, ≥ 1:28 | 163 | 170 | 74
  Month 6, ≥ 1:56: number analyzed (Participants) | 163 | 0 | 0
  Month 6, ≥ 1:56 | 158 | 0 | 0
  Month 12, ≥ 1:56: number analyzed (Participants) | 75 | 164 | 0
  Month 12, ≥ 1:56 | 74 | 155 | 0
  Month 24, ≥ 1:56: number analyzed (Participants) | 75 | 75 | 75
  Month 24, ≥ 1:56 | 60 | 71 | 29
  Month 36, ≥ 1:56: number analyzed (Participants) | 75 | 74 | 75
  Month 36, ≥ 1:56 | 52 | 60 | 27
  Month 48, ≥ 1:56: number analyzed (Participants) | 75 | 75 | 75
  Month 48, ≥ 1:56 | 65 | 65 | 74
  Month 6/12/36 + 21 days, ≥ 1:56: number analyzed (Participants) | 163 | 170 | 74
  Month 6/12/36 + 21 days, ≥ 1:56 | 163 | 170 | 74
  Month 6, ≥ 1:112: number analyzed (Participants) | 163 | 0 | 0
  Month 6, ≥ 1:112 | 134 | 0 | 0
  Month 12, ≥ 1:112: number analyzed (Participants) | 75 | 164 | 0
  Month 12, ≥ 1:112 | 59 | 137 | 0
  Month 24, ≥ 1:112: number analyzed (Participants) | 75 | 75 | 75
  Month 24, ≥ 1:112 | 34 | 50 | 6
  Month 36, ≥ 1:112: number analyzed (Participants) | 75 | 74 | 75
  Month 36, ≥ 1:112 | 30 | 43 | 5
  Month 48, ≥ 1:112: number analyzed (Participants) | 75 | 75 | 75
  Month 48, ≥ 1:112 | 30 | 48 | 68
  Month 6/12/36 + 21 days, ≥ 1:112: number analyzed (Participants) | 163 | 170 | 74
  Month 6/12/36 + 21 days, ≥ 1:112 | 163 | 170 | 72

24. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms
Description: Assessed solicited local symptoms were ecchymosis, induration, pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = pain that prevented normal activity. Grade 3 ecchymosis/induration/redness/swelling = redness/swelling spreading beyond 100 millimeters (mm) of injection site.
Time Frame: During the 7-day (Days 0-6) post-vaccination period - subjects boosted at Month 12 and Month 36
Population: The analysis was performed on the Total Vaccinated cohort, which included all booster-vaccinated subjects for whom data were available and who had their symptom sheets filled in.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A M12 Group | GSK1562902A M36 Group
Number analyzed (Participants) | 188 | 386
Participants
  Any Ecchymosis | 2 | 1
  Grade 3 Ecchymosis | 0 | 0
  Any Induration | 17 | 23
  Grade 3 Induration | 0 | 0
  Any Pain | 158 | 306
  Grade 3 Pain | 11 | 17
  Any Redness | 13 | 28
  Grade 3 Redness | 0 | 0
  Any Swelling | 23 | 44
  Grade 3 Swelling | 0 | 0

25. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptom
Description: Assessed solicited general symptoms were arthralgia, fatigue, headache, myalgia, shivering, sweating and fever [defined as axillary temperature equal to or above (≥) 38 degrees Celsius (°C)]. Any = occurrence of the symptom regardless of intensity grade. Grade 3 symptom = symptom that prevented normal activity. Grade 3 fever = fever ≥ 39.0 °C. Related = symptom assessed by the investigator as causally related to the study vaccination.
Time Frame: During the 7-day (Days 0-6) post-vaccination period - subjects boosted at Month 12 and 36
Population: The analysis was performed on the Total Vaccinated cohort, which included all booster-vaccinated subjects for whom data were available and who has their symptom sheets filled in.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A M12 Group | GSK1562902A M36 Group
Number analyzed (Participants) | 188 | 386
Participants
  Any Arthralgia | 48 | 99
  Grade 3 Arthralgia | 6 | 7
  Related Arthralgia | 45 | 95
  Any Fatigue | 112 | 216
  Grade 3 Fatigue | 12 | 19
  Related Fatigue | 105 | 213
  Any Headache | 76 | 138
  Grade 3 Headache | 12 | 7
  Related Headache | 69 | 134
  Any Myalgia | 123 | 235
  Grade 3 Myalgia | 14 | 17
  Related Myalgia | 119 | 226
  Any Shivering | 26 | 51
  Grade 3 Shivering | 3 | 8
  Related Shivering | 26 | 49
  Any Sweating | 22 | 54
  Grade 3 Sweating | 0 | 2
  Related Sweating | 20 | 52
  Any Temperature | 15 | 24
  Grade 3 Temperature | 1 | 3
  Related Temperature | 14 | 23

26. Secondary Outcome: Number of Subjects With Adverse Events of Specific Interest (AESIs)
Description: An AESI was defined as an AE including autoimmune diseases and other mediated inflammatory disorders and assessed by the investigator as specific to the treatment administration.
Time Frame: During the entire study period (From Month 12 to Month 48)
Population: The analysis was performed on the Total Vaccinated cohort, which included all booster-vaccinated subjects for whom data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A M6 Group | GSK1562902A M12 Group | GSK1562902A M36 Group
Number analyzed (Participants) | 196 | 170 | 367
Participants | 0 | 0 | 1

27. Secondary Outcome: Frequency of Antigen-specific CD4 T-cells (Per 10E6) in Tests Identified as Producing at Least Two Out of Four Different Cytokines (for A/Indonesia/05/2005 Strain)
Description: Among cytokines expressed after background reduction were cluster of differentiation 4 all doubles (CD4 all doubles), cluster of differentiation 40-ligand (CD40-L), interferon-gamma (IFN-γ), interleukin-2 (IL-2) and tumour necrosis factor-alpha (TNF-α). The flu strain assessed was H5N1 A/Indonesia/05/2005.
Time Frame: At Months 6, 12, 18, 24, 30, 36, 42 and 48 and at Months 6/12/36 + 21 days
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: T-cells/million cells
Arm/Group | GSK1562902A M6 Group | GSK1562902A M12 Group | GSK1562902A M36 Group
Number analyzed (Participants) | 5 | 7 | 15
T-cells/million cells
  CD4-All doubles, Month 6: number analyzed (Participants) | 2 | 3 | 4
  CD4-All doubles, Month 6 | 1119.00 [895.00 to 1343.00] | 1862.00 [1836.00 to 2980.00] | 3109.50 [2851.50 to 3576.50]
  CD4-All doubles, Month 12: number analyzed (Participants) | 5 | 7 | 13
  CD4-All doubles, Month 12 | 2620.00 [2422.00 to 2935.00] | 1599.00 [1438.00 to 1929.00] | 1443.00 [1065.00 to 2070.00]
  CD4-All doubles, Month 18 | 2060.00 [1611.00 to 2263.00] | 2335.00 [1820.00 to 4476.00] | 1590.00 [1232.00 to 2010.00]
  CD4-All doubles, Month 24: number analyzed (Participants) | 4 | 5 | 13
  CD4-All doubles, Month 24 | 2565.50 [1890.50 to 3120.00] | 3517.00 [1840.00 to 4567.00] | 1396.00 [1259.00 to 1684.00]
  CD4-All doubles, Month 30: number analyzed (Participants) | 2 | 5 | 13
  CD4-All doubles, Month 30 | 3147.50 [2539.00 to 3756.00] | 3907.00 [1281.00 to 4371.00] | 1670.00 [1126.00 to 2256.00]
  CD4-All doubles, Month 36: number analyzed (Participants) | 4 | 7 | 13
  CD4-All doubles, Month 36 | 1689.50 [839.00 to 2649.00] | 2506.00 [962.00 to 3842.00] | 995.00 [849.00 to 1291.00]
  CD4-All doubles, Month 42 | 1656.00 [877.00 to 2734.00] | 2311.00 [1068.00 to 3328.00] | 2129.00 [1597.00 to 2475.00]
  CD4-All doubles, Month 48: number analyzed (Participants) | 5 | 6 | 13
  CD4-All doubles, Month 48 | 1496.00 [1309.00 to 1878.00] | 2054.50 [1404.00 to 4027.00] | 2064.00 [1479.00 to 2906.00]
  CD4-All doubles, Month 6/12/36 + 21 days: number analyzed (Participants) | 4 | 6 | 12
  CD4-All doubles, Month 6/12/36 + 21 days | 5401.50 [3071.00 to 8338.50] | 9553.00 [4183.00 to 17658.00] | 5057.00 [4388.00 to 7039.00]
  CD4-CD40L, Month 6: number analyzed (Participants) | 2 | 3 | 4
  CD4-CD40L, Month 6 | 1045.00 [817.00 to 1273.00] | 1792.00 [1691.00 to 2986.00] | 2829.50 [2605.50 to 3232.00]
  CD4-CD40L, Month 12: number analyzed (Participants) | 5 | 7 | 13
  CD4-CD40L, Month 12 | 2634.00 [2382.00 to 2917.00] | 1494.00 [1425.00 to 1872.00] | 1372.00 [1039.00 to 1991.00]
  CD4-CD40L, Month 18 | 2025.00 [1609.00 to 2223.00] | 2240.00 [1692.00 to 4454.00] | 1518.00 [1148.00 to 1929.00]
  CD4-CD40L, Month 24: number analyzed (Participants) | 4 | 5 | 13
  CD4-CD40L, Month 24 | 2583.00 [1857.00 to 3135.50] | 3435.00 [1801.00 to 4486.00] | 1395.00 [1240.00 to 1724.00]
  CD4-CD40L, Month 30: number analyzed (Participants) | 2 | 5 | 13
  CD4-CD40L, Month 30 | 3113.00 [2497.00 to 3729.00] | 3652.00 [1296.00 to 4172.00] | 1685.00 [1153.00 to 2195.00]
  CD4-CD40L, Month 36: number analyzed (Participants) | 4 | 7 | 13
  CD4-CD40L, Month 36 | 1683.00 [848.00 to 2642.50] | 2453.00 [958.00 to 3867.00] | 975.00 [849.00 to 1278.00]
  CD4-CD40L, Month 42 | 1656.00 [873.00 to 2719.00] | 2243.00 [1055.00 to 3311.00] | 2142.00 [1584.00 to 2451.00]
  CD4-CD40L, Month 48: number analyzed (Participants) | 5 | 6 | 13
  CD4-CD40L, Month 48 | 1496.00 [1252.00 to 1799.00] | 2013.50 [1418.00 to 3905.00] | 2008.00 [1433.00 to 2856.00]
  CD4-CD40L, Month 6/12/36 + 21 days: number analyzed (Participants) | 4 | 6 | 12
  CD4-CD40L, Month 6/12/36 + 21 days | 5292.00 [3027.00 to 8110.00] | 9416.00 [4129.00 to 17348.00] | 5038.00 [4283.00 to 7018.00]
  CD4-IFN-γ, Month 6: number analyzed (Participants) | 2 | 3 | 4
  CD4-IFN-γ, Month 6 | 537.50 [431.00 to 644.00] | 1189.00 [862.00 to 1570.00] | 2134.00 [1755.50 to 2525.50]
  CD4-IFN-γ, Month 12: number analyzed (Participants) | 5 | 7 | 13
  CD4-IFN-γ, Month 12 | 1217.00 [1046.00 to 1782.00] | 994.00 [607.00 to 1073.00] | 852.00 [525.00 to 1081.00]
  CD4-IFN-γ, Month 18 | 989.00 [956.00 to 1206.00] | 1306.00 [1049.00 to 2032.00] | 959.00 [678.00 to 1151.00]
  CD4-IFN-γ, Month 24: number analyzed (Participants) | 4 | 5 | 13
  CD4-IFN-γ, Month 24 | 1590.50 [1036.00 to 1905.00] | 2036.00 [854.00 to 2315.00] | 787.00 [655.00 to 947.00]
  CD4-IFN-γ, Month 30: number analyzed (Participants) | 2 | 5 | 13
  CD4-IFN-γ, Month 30 | 1829.00 [1464.00 to 2194.00] | 1892.00 [838.00 to 2466.00] | 1096.00 [758.00 to 1330.00]
  CD4-IFN-γ, Month 36: number analyzed (Participants) | 4 | 7 | 13
  CD4-IFN-γ, Month 36 | 1026.00 [481.00 to 1548.50] | 1452.00 [606.00 to 2023.00] | 543.00 [380.00 to 662.00]
  CD4-IFN-γ, Month 42 | 698.00 [349.00 to 1416.00] | 1336.00 [568.00 to 1805.00] | 1119.00 [714.00 to 1728.00]
  CD4-IFN-γ, Month 48: number analyzed (Participants) | 5 | 6 | 13
  CD4-IFN-γ, Month 48 | 964.00 [721.00 to 1157.00] | 1085.00 [787.00 to 2692.00] | 1334.00 [553.00 to 1822.00]
  CD4-IFN-γ, Month 6/12/36 + 21 days: number analyzed (Participants) | 4 | 6 | 12
  CD4-IFN-γ, Month 6/12/36 + 21 days | 3255.00 [1676.00 to 4878.50] | 4661.50 [1676.00 to 11231.00] | 2077.50 [1745.00 to 2972.50]
  CD4-IL-2, Month 6: number analyzed (Participants) | 2 | 3 | 4
  CD4-IL-2, Month 6 | 883.50 [612.00 to 1155.00] | 1657.00 [1639.00 to 2798.00] | 2799.00 [2495.50 to 3049.00]
  CD4-IL-2, Month 12: number analyzed (Participants) | 5 | 7 | 13
  CD4-IL-2, Month 12 | 2580.00 [2290.00 to 2770.00] | 1649.00 [1293.00 to 1865.00] | 1335.00 [961.00 to 1859.00]
  CD4-IL-2, Month 18 | 1990.00 [1430.00 to 2290.00] | 2297.00 [1694.00 to 4071.00] | 1224.00 [1164.00 to 1695.00]
  CD4-IL-2, Month 24: number analyzed (Participants) | 4 | 5 | 13
  CD4-IL-2, Month 24 | 2423.50 [1653.50 to 2937.00] | 3256.00 [1653.00 to 4370.00] | 1187.00 [1107.00 to 1534.00]
  CD4-IL-2, Month 30: number analyzed (Participants) | 2 | 5 | 13
  CD4-IL-2, Month 30 | 2830.50 [2319.00 to 3342.00] | 3459.00 [1251.00 to 4078.00] | 1506.00 [1037.00 to 2122.00]
  CD4-IL-2, Month 36: number analyzed (Participants) | 4 | 7 | 13
  CD4-IL-2, Month 36 | 1490.50 [770.00 to 2396.00] | 2247.00 [1015.00 to 3681.00] | 846.00 [755.00 to 1077.00]
  CD4-IL-2, Month 42 | 1533.00 [801.00 to 2472.00] | 2123.00 [1069.00 to 3248.00] | 2072.00 [1472.00 to 2250.00]
  CD4-IL-2, Month 48: number analyzed (Participants) | 5 | 6 | 13
  CD4-IL-2, Month 48 | 1373.00 [1115.00 to 1814.00] | 1906.00 [1264.00 to 3659.00] | 1926.00 [1292.00 to 2721.00]
  CD4-IL-2, Month 6/12/36 + 21 days: number analyzed (Participants) | 4 | 6 | 12
  CD4-IL-2, Month 6/12/36 + 21 days | 4972.50 [2846.00 to 7782.50] | 8993.00 [3979.00 to 16403.00] | 4532.00 [4133.50 to 6494.00]
  CD4-TNF-α, Month 6: number analyzed (Participants) | 2 | 3 | 4
  CD4-TNF-α, Month 6 | 909.00 [649.00 to 1169.00] | 1644.00 [1334.00 to 2617.00] | 2579.00 [2327.00 to 2985.50]
  CD4-TNF-α, Month 12: number analyzed (Participants) | 5 | 7 | 13
  CD4-TNF-α, Month 12 | 2528.00 [2107.00 to 2752.00] | 1515.00 [1346.00 to 1674.00] | 1174.00 [975.00 to 2031.00]
  CD4-TNF-α, Month 18 | 1462.00 [1459.00 to 1585.00] | 1810.00 [1451.00 to 3453.00] | 1160.00 [894.00 to 1492.00]
  CD4-TNF-α, Month 24: number analyzed (Participants) | 4 | 5 | 13
  CD4-TNF-α, Month 24 | 2084.50 [1331.50 to 2414.50] | 2972.00 [1281.00 to 4109.00] | 1107.00 [1005.00 to 1333.00]
  CD4-TNF-α, Month 30: number analyzed (Participants) | 2 | 5 | 13
  CD4-TNF-α, Month 30 | 2442.50 [2119.00 to 2766.00] | 3247.00 [1042.00 to 3614.00] | 1269.00 [1036.00 to 1889.00]
  CD4-TNF-α, Month 36: number analyzed (Participants) | 4 | 7 | 13
  CD4-TNF-α, Month 36 | 1476.50 [697.50 to 2289.00] | 2291.00 [951.00 to 3523.00] | 917.00 [640.00 to 969.00]
  CD4-TNF-α, Month 42 | 1218.00 [558.00 to 2068.00] | 1901.00 [811.00 to 2695.00] | 1675.00 [1218.00 to 2018.00]
  CD4-TNF-α, Month 48: number analyzed (Participants) | 5 | 6 | 13
  CD4-TNF-α, Month 48 | 1169.00 [1028.00 to 1376.00] | 1769.50 [1166.00 to 3244.00] | 1794.00 [1106.00 to 2505.00]
  CD4-TNF-α, Month 6/12/36 + 21 days: number analyzed (Participants) | 4 | 6 | 12
  CD4-TNF-α, Month 6/12/36 + 21 days | 4249.50 [2151.50 to 6892.00] | 8466.00 [3885.00 to 17018.00] | 3726.50 [3454.50 to 5939.50]

28. Secondary Outcome: Frequency of Antigen-specific CD4 T-cells (Per 10E6) in Tests Identified as Producing at Least Two Out of Four Different Cytokines (for A/Vietnam/1194/2004 Strain)
Description: Among cytokines expressed after background reduction were cluster of differentiation 4 all doubles (CD4 all doubles), cluster of differentiation 40-ligand (CD40-L), interferon-gamma (IFN-γ), interleukin-2 (IL-2) and tumour necrosis factor-alpha (TNF-α). The flu strain assessed was H5N1 A/Vietnam/1194/2004.
Time Frame: At Months 6, 12, 18, 24, 30, 36, 42 and 48 and at Months 6/12/36 + 21 days
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: T-cells/million cells
Arm/Group | GSK1562902A M6 Group | GSK1562902A M12 Group | GSK1562902A M36 Group
Number analyzed (Participants) | 5 | 7 | 15
T-cells/million cells
  CD4-All doubles, Month 6: number analyzed (Participants) | 2 | 3 | 8
  CD4-All doubles, Month 6 | 1615.50 [918.00 to 2313.00] | 2133.00 [1392.00 to 2727.00] | 3047.00 [1913.00 to 3790.00]
  CD4-All doubles, Month 12: number analyzed (Participants) | 5 | 7 | 14
  CD4-All doubles, Month 12 | 2410.00 [2288.00 to 3872.00] | 1889.00 [1263.00 to 2305.00] | 1849.50 [1327.00 to 2605.00]
  CD4-All doubles, Month 18 | 2505.00 [2491.00 to 2790.00] | 4073.00 [2335.00 to 4833.00] | 1658.00 [1301.00 to 1927.00]
  CD4-All doubles, Month 24: number analyzed (Participants) | 4 | 5 | 13
  CD4-All doubles, Month 24 | 2720.00 [1726.50 to 3263.50] | 3945.00 [1666.00 to 4592.00] | 1472.00 [1264.00 to 1906.00]
  CD4-All doubles, Month 30: number analyzed (Participants) | 2 | 5 | 13
  CD4-All doubles, Month 30 | 2959.50 [2252.00 to 3667.00] | 3713.00 [1996.00 to 5220.00] | 1478.00 [1275.00 to 2210.00]
  CD4-All doubles, Month 36: number analyzed (Participants) | 4 | 7 | 13
  CD4-All doubles, Month 36 | 1420.00 [645.00 to 2468.00] | 2149.00 [977.00 to 4081.00] | 1097.00 [836.00 to 1395.00]
  CD4-All doubles, Month 42 | 1354.00 [1190.00 to 2571.00] | 2264.00 [1157.00 to 3817.00] | 2555.00 [1665.00 to 2882.00]
  CD4-All doubles, Month 48: number analyzed (Participants) | 5 | 6 | 13
  CD4-All doubles, Month 48 | 1600.00 [1374.00 to 2493.00] | 2087.50 [1236.00 to 4476.00] | 2332.00 [1451.00 to 3052.00]
  CD4-All doubles, Month 6/12/36 + 21 days: number analyzed (Participants) | 4 | 6 | 12
  CD4-All doubles, Month 6/12/36 + 21 days | 7067.50 [3359.50 to 10769.50] | 10061.50 [4553.00 to 18155.00] | 5315.50 [4283.50 to 7167.00]
  CD4-CD40L, Month 6: number analyzed (Participants) | 2 | 3 | 8
  CD4-CD40L, Month 6 | 1586.00 [857.00 to 2315.00] | 1998.00 [1335.00 to 2496.00] | 2937.50 [1851.00 to 3612.00]
  CD4-CD40L, Month 12: number analyzed (Participants) | 5 | 7 | 14
  CD4-CD40L, Month 12 | 2384.00 [2257.00 to 3832.00] | 1863.00 [1206.00 to 2249.00] | 1741.50 [1327.00 to 2484.00]
  CD4-CD40L, Month 18 | 2517.00 [2456.00 to 2776.00] | 3980.00 [2294.00 to 4803.00] | 1607.00 [1274.00 to 1819.00]
  CD4-CD40L, Month 24: number analyzed (Participants) | 4 | 5 | 13
  CD4-CD40L, Month 24 | 2735.50 [1693.00 to 3280.50] | 3932.00 [1667.00 to 4539.00] | 1490.00 [1279.00 to 1933.00]
  CD4-CD40L, Month 30: number analyzed (Participants) | 2 | 5 | 13
  CD4-CD40L, Month 30 | 2882.00 [2175.00 to 3589.00] | 3607.00 [1908.00 to 5200.00] | 1449.00 [1289.00 to 2123.00]
  CD4-CD40L, Month 36: number analyzed (Participants) | 4 | 7 | 13
  CD4-CD40L, Month 36 | 1406.00 [654.00 to 2475.00] | 2122.00 [962.00 to 4049.00] | 1098.00 [783.00 to 1328.00]
  CD4-CD40L, Month 42 | 1340.00 [1174.00 to 2557.00] | 2265.00 [1116.00 to 3800.00] | 2502.00 [1638.00 to 2868.00]
  CD4-CD40L, Month 48: number analyzed (Participants) | 5 | 6 | 13
  CD4-CD40L, Month 48 | 1618.00 [1387.00 to 2449.00] | 2008.50 [1236.00 to 4383.00] | 2332.00 [1451.00 to 2885.00]
  CD4-CD40L, Month 6/12/36 + 21 days: number analyzed (Participants) | 4 | 6 | 12
  CD4-CD40L, Month 6/12/36 + 21 days | 6931.00 [3256.00 to 10610.50] | 9587.00 [4451.00 to 17713.00] | 5296.00 [4267.00 to 7144.50]
  CD4-IFN-γ, Month 6: number analyzed (Participants) | 2 | 3 | 8
  CD4-IFN-γ, Month 6 | 826.00 [365.00 to 1287.00] | 999.00 [452.00 to 1623.00] | 1420.00 [948.00 to 2423.00]
  CD4-IFN-γ, Month 12: number analyzed (Participants) | 5 | 7 | 14
  CD4-IFN-γ, Month 12 | 1108.00 [876.00 to 2433.00] | 884.00 [608.00 to 925.00] | 869.50 [633.00 to 1329.00]
  CD4-IFN-γ, Month 18 | 1395.00 [1047.00 to 1573.00] | 1927.00 [1061.00 to 2642.00] | 941.00 [548.00 to 1263.00]
  CD4-IFN-γ, Month 24: number analyzed (Participants) | 4 | 5 | 13
  CD4-IFN-γ, Month 24 | 1659.00 [1046.00 to 1846.00] | 2439.00 [613.00 to 2625.00] | 847.00 [658.00 to 1112.00]
  CD4-IFN-γ, Month 30: number analyzed (Participants) | 2 | 5 | 13
  CD4-IFN-γ, Month 30 | 1885.50 [1473.00 to 2298.00] | 2248.00 [1264.00 to 2469.00] | 1074.00 [859.00 to 1155.00]
  CD4-IFN-γ, Month 36: number analyzed (Participants) | 4 | 7 | 13
  CD4-IFN-γ, Month 36 | 813.50 [436.00 to 1244.00] | 1260.00 [512.00 to 2163.00] | 621.00 [526.00 to 730.00]
  CD4-IFN-γ, Month 42 | 547.00 [546.00 to 1515.00] | 1218.00 [449.00 to 2058.00] | 1228.00 [949.00 to 1682.00]
  CD4-IFN-γ, Month 48: number analyzed (Participants) | 5 | 6 | 13
  CD4-IFN-γ, Month 48 | 749.00 [697.00 to 1682.00] | 1007.00 [646.00 to 2797.00] | 1223.00 [658.00 to 1866.00]
  CD4-IFN-γ, Month 6/12/36 + 21 days: number analyzed (Participants) | 4 | 6 | 12
  CD4-IFN-γ, Month 6/12/36 + 21 days | 3608.50 [1467.50 to 5510.50] | 4918.00 [1852.00 to 9857.00] | 2142.00 [1763.50 to 2954.50]
  CD4-IL-2, Month 6: number analyzed (Participants) | 2 | 3 | 8
  CD4-IL-2, Month 6 | 1493.00 [952.00 to 2034.00] | 1957.00 [1382.00 to 2522.00] | 2910.50 [1768.50 to 3368.50]
  CD4-IL-2, Month 12: number analyzed (Participants) | 5 | 7 | 14
  CD4-IL-2, Month 12 | 2305.00 [2075.00 to 3663.00] | 1729.00 [1286.00 to 2197.00] | 1759.00 [1393.00 to 2469.00]
  CD4-IL-2, Month 18 | 2431.00 [2425.00 to 2750.00] | 4073.00 [2281.00 to 4495.00] | 1592.00 [1235.00 to 1833.00]
  CD4-IL-2, Month 24: number analyzed (Participants) | 4 | 5 | 13
  CD4-IL-2, Month 24 | 2598.00 [1545.50 to 3129.50] | 3799.00 [1480.00 to 4419.00] | 1454.00 [1093.00 to 1693.00]
  CD4-IL-2, Month 30: number analyzed (Participants) | 2 | 5 | 13
  CD4-IL-2, Month 30 | 2773.00 [2137.00 to 3409.00] | 3537.00 [1910.00 to 5234.00] | 1344.00 [1262.00 to 2086.00]
  CD4-IL-2, Month 36: number analyzed (Participants) | 4 | 7 | 13
  CD4-IL-2, Month 36 | 1301.00 [674.50 to 2268.00] | 2240.00 [798.00 to 3945.00] | 891.00 [808.00 to 1247.00]
  CD4-IL-2, Month 42 | 1218.00 [1125.00 to 2362.00] | 2179.00 [1075.00 to 3878.00] | 2323.00 [1693.00 to 2676.00]
  CD4-IL-2, Month 48: number analyzed (Participants) | 5 | 6 | 13
  CD4-IL-2, Month 48 | 1169.00 [966.00 to 2422.00] | 1931.50 [1151.00 to 3830.00] | 2218.00 [1271.00 to 2642.00]
  CD4-IL-2, Month 6/12/36 + 21 days: number analyzed (Participants) | 4 | 6 | 12
  CD4-IL-2, Month 6/12/36 + 21 days | 6557.00 [3110.50 to 9871.00] | 9252.00 [4333.00 to 17247.00] | 4759.50 [3940.50 to 6757.00]
  CD4-TNF-α, Month 6: number analyzed (Participants) | 2 | 3 | 8
  CD4-TNF-α, Month 6 | 1280.50 [803.00 to 1758.00] | 1768.00 [1240.00 to 1938.00] | 2540.00 [1451.50 to 2899.00]
  CD4-TNF-α, Month 12: number analyzed (Participants) | 5 | 7 | 14
  CD4-TNF-α, Month 12 | 1784.00 [1683.00 to 3353.00] | 1488.00 [925.00 to 1636.00] | 1404.00 [1142.00 to 2111.00]
  CD4-TNF-α, Month 18 | 2258.00 [2147.00 to 2346.00] | 3357.00 [1879.00 to 4452.00] | 1392.00 [996.00 to 1518.00]
  CD4-TNF-α, Month 24: number analyzed (Participants) | 4 | 5 | 13
  CD4-TNF-α, Month 24 | 1871.00 [1145.50 to 2420.00] | 3252.00 [1107.00 to 4049.00] | 1131.00 [934.00 to 1419.00]
  CD4-TNF-α, Month 30: number analyzed (Participants) | 2 | 5 | 13
  CD4-TNF-α, Month 30 | 2191.00 [1720.00 to 2662.00] | 3246.00 [1438.00 to 4397.00] | 1246.00 [987.00 to 1662.00]
  CD4-TNF-α, Month 36: number analyzed (Participants) | 4 | 7 | 13
  CD4-TNF-α, Month 36 | 1145.00 [501.00 to 1974.00] | 1935.00 [820.00 to 3658.00] | 829.00 [569.00 to 1071.00]
  CD4-TNF-α, Month 42 | 1094.00 [818.00 to 2000.00] | 1819.00 [858.00 to 3069.00] | 1863.00 [1390.00 to 2182.00]
  CD4-TNF-α, Month 48: number analyzed (Participants) | 5 | 6 | 13
  CD4-TNF-α, Month 48 | 1376.00 [1197.00 to 1769.00] | 1737.00 [941.00 to 3622.00] | 1781.00 [1203.00 to 2307.00]
  CD4-TNF-α, Month 6/12/36 + 21 days: number analyzed (Participants) | 4 | 6 | 12
  CD4-TNF-α, Month 6/12/36 + 21 days | 5527.50 [2298.00 to 8633.50] | 7385.50 [3438.00 to 16134.00] | 3899.00 [3218.00 to 6044.50]

29. Secondary Outcome: Frequency of Antigen-specific CD8 T-cells (Per 10E6) in Tests Identified as Producing at Least Two Out of Four Different Cytokines (for A/Indonesia/05/2005 Strain)
Description: Among cytokines expressed after background reduction were cluster of differentiation 8 all doubles (CD8 all doubles), cluster of differentiation 40-ligand (CD40-L), interleukin-2 (IL-2), interferon-gamma (IFN-γ) and tumour necrosis factor-alpha (TNF-α). The flu strain assessed was H5N1 A/Indonesia/05/2005.
Time Frame: At Months 6, 12, 18, 24, 30, 36, 42 and 48 and at Months 6/12/36 + 21 days
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: T-cells/million cells
Arm/Group | GSK1562902A M6 Group | GSK1562902A M12 Group | GSK1562902A M36 Group
Number analyzed (Participants) | 5 | 7 | 15
T-cells/million cells
  CD8-All doubles, Month 6: number analyzed (Participants) | 2 | 3 | 4
  CD8-All doubles, Month 6 | 34.50 [26.00 to 43.00] | 1.00 [1.00 to 42.00] | 14.00 [7.00 to 48.00]
  CD8-All doubles, Month 12: number analyzed (Participants) | 5 | 7 | 13
  CD8-All doubles, Month 12 | 1.00 [1.00 to 4.00] | 26.00 [1.00 to 111.00] | 44.00 [1.00 to 141.00]
  CD8-All doubles, Month 18: number analyzed (Participants) | 5 | 7 | 14
  CD8-All doubles, Month 18 | 1.00 [1.00 to 1.00] | 120.00 [27.00 to 139.00] | 27.00 [1.00 to 220.00]
  CD8-All doubles, Month 24: number analyzed (Participants) | 4 | 5 | 13
  CD8-All doubles, Month 24 | 23.00 [1.00 to 73.00] | 51.00 [1.00 to 134.00] | 88.00 [41.00 to 208.00]
  CD8-All doubles, Month 30: number analyzed (Participants) | 2 | 5 | 13
  CD8-All doubles, Month 30 | 2.50 [1.00 to 4.00] | 1.00 [1.00 to 2.00] | 37.00 [1.00 to 47.00]
  CD8-All doubles, Month 36: number analyzed (Participants) | 4 | 7 | 13
  CD8-All doubles, Month 36 | 38.50 [14.00 to 52.00] | 17.00 [1.00 to 78.00] | 35.00 [1.00 to 77.00]
  CD8-All doubles, Month 42 | 19.00 [1.00 to 23.00] | 3.00 [1.00 to 24.00] | 1.00 [1.00 to 42.00]
  CD8-All doubles, Month 48: number analyzed (Participants) | 5 | 6 | 13
  CD8-All doubles, Month 48 | 30.00 [1.00 to 59.00] | 20.50 [1.00 to 86.00] | 1.00 [1.00 to 60.00]
  CD8-All doubles, Month 6/12/36 + 21 days: number analyzed (Participants) | 4 | 6 | 12
  CD8-All doubles, Month 6/12/36 + 21 days | 73.00 [26.50 to 130.50] | 159.50 [93.00 to 217.00] | 45.50 [22.50 to 101.00]
  CD8-CD40L, Month 6: number analyzed (Participants) | 2 | 3 | 4
  CD8-CD40L, Month 6 | 34.00 [25.00 to 43.00] | 1.00 [1.00 to 68.00] | 3.50 [1.00 to 8.50]
  CD8-CD40L, Month 12: number analyzed (Participants) | 5 | 7 | 13
  CD8-CD40L, Month 12 | 1.00 [1.00 to 95.00] | 1.00 [1.00 to 111.00] | 1.00 [1.00 to 75.00]
  CD8-CD40L, Month 18: number analyzed (Participants) | 5 | 7 | 14
  CD8-CD40L, Month 18 | 1.00 [1.00 to 1.00] | 9.00 [1.00 to 36.00] | 1.00 [1.00 to 22.00]
  CD8-CD40L, Month 24: number analyzed (Participants) | 4 | 5 | 13
  CD8-CD40L, Month 24 | 55.50 [8.50 to 112.00] | 32.00 [26.00 to 35.00] | 61.00 [1.00 to 91.00]
  CD8-CD40L, Month 30: number analyzed (Participants) | 2 | 5 | 13
  CD8-CD40L, Month 30 | 3.00 [1.00 to 5.00] | 1.00 [1.00 to 3.00] | 1.00 [1.00 to 16.00]
  CD8-CD40L, Month 36: number analyzed (Participants) | 4 | 7 | 13
  CD8-CD40L, Month 36 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 19.00] | 1.00 [1.00 to 20.00]
  CD8-CD40L, Month 42 | 1.00 [1.00 to 9.00] | 1.00 [1.00 to 13.00] | 1.00 [1.00 to 1.00]
  CD8-CD40L, Month 48: number analyzed (Participants) | 5 | 6 | 13
  CD8-CD40L, Month 48 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 3.00]
  CD8-CD40L, Month 6/12/36 + 21 days: number analyzed (Participants) | 4 | 6 | 15
  CD8-CD40L, Month 6/12/36 + 21 days | 78.50 [39.00 to 96.50] | 28.00 [1.00 to 102.00] | 30.50 [1.00 to 41.50]
  CD8-IFN-γ, Month 6: number analyzed (Participants) | 2 | 3 | 4
  CD8-IFN-γ, Month 6 | 22.00 [1.00 to 43.00] | 1.00 [1.00 to 42.00] | 8.00 [1.00 to 48.00]
  CD8-IFN-γ, Month 12: number analyzed (Participants) | 5 | 7 | 13
  CD8-IFN-γ, Month 12 | 1.00 [1.00 to 44.00] | 54.00 [1.00 to 86.00] | 1.00 [1.00 to 91.00]
  CD8-IFN-γ, Month 18: number analyzed (Participants) | 5 | 7 | 14
  CD8-IFN-γ, Month 18 | 1.00 [1.00 to 3.00] | 120.00 [36.00 to 139.00] | 27.00 [1.00 to 220.00]
  CD8-IFN-γ, Month 24: number analyzed (Participants) | 4 | 5 | 13
  CD8-IFN-γ, Month 24 | 23.00 [1.00 to 55.50] | 30.00 [1.00 to 117.00] | 95.00 [41.00 to 142.00]
  CD8-IFN-γ, Month 30: number analyzed (Participants) | 2 | 5 | 13
  CD8-IFN-γ, Month 30 | 2.50 [1.00 to 4.00] | 1.00 [1.00 to 2.00] | 18.00 [1.00 to 26.00]
  CD8-IFN-γ, Month 36: number analyzed (Participants) | 4 | 7 | 13
  CD8-IFN-γ, Month 36 | 38.50 [19.00 to 52.00] | 25.00 [3.00 to 39.00] | 20.00 [1.00 to 77.00]
  CD8-IFN-γ, Month 42 | 1.00 [1.00 to 9.00] | 1.00 [1.00 to 3.00] | 1.00 [1.00 to 27.00]
  CD8-IFN-γ, Month 48: number analyzed (Participants) | 5 | 6 | 13
  CD8-IFN-γ, Month 48 | 1.00 [1.00 to 1.00] | 29.00 [1.00 to 86.00] | 1.00 [1.00 to 60.00]
  CD8-IFN-γ, Month 6/12/36 + 21 days: number analyzed (Participants) | 4 | 6 | 15
  CD8-IFN-γ, Month 6/12/36 + 21 days | 59.50 [26.50 to 117.00] | 93.50 [1.00 to 165.00] | 35.00 [1.00 to 65.50]
  CD8-IL-2, Month 6: number analyzed (Participants) | 2 | 3 | 4
  CD8-IL-2, Month 6 | 12.50 [1.00 to 24.00] | 1.00 [1.00 to 34.00] | 32.00 [16.00 to 36.50]
  CD8-IL-2, Month 12: number analyzed (Participants) | 5 | 7 | 13
  CD8-IL-2, Month 12 | 1.00 [1.00 to 47.00] | 1.00 [1.00 to 27.00] | 31.00 [1.00 to 184.00]
  CD8-IL-2, Month 18: number analyzed (Participants) | 5 | 7 | 14
  CD8-IL-2, Month 18 | 1.00 [1.00 to 1.00] | 47.00 [9.00 to 78.00] | 27.50 [1.00 to 161.00]
  CD8-IL-2, Month 24: number analyzed (Participants) | 4 | 5 | 13
  CD8-IL-2, Month 24 | 5.00 [1.00 to 13.50] | 1.00 [1.00 to 19.00] | 39.00 [24.00 to 60.00]
  CD8-IL-2, Month 30: number analyzed (Participants) | 2 | 5 | 13
  CD8-IL-2, Month 30 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 3.00] | 16.00 [1.00 to 36.00]
  CD8-IL-2, Month 36: number analyzed (Participants) | 4 | 7 | 13
  CD8-IL-2, Month 36 | 38.50 [14.00 to 52.00] | 17.00 [1.00 to 58.00] | 20.00 [1.00 to 38.00]
  CD8-IL-2, Month 42 | 19.00 [1.00 to 23.00] | 13.00 [1.00 to 24.00] | 1.00 [1.00 to 42.00]
  CD8-IL-2, Month 48: number analyzed (Participants) | 5 | 6 | 13
  CD8-IL-2, Month 48 | 30.00 [1.00 to 55.00] | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 44.00]
  CD8-IL-2, Month 6/12/36 + 21 days: number analyzed (Participants) | 4 | 6 | 12
  CD8-IL-2, Month 6/12/36 + 21 days | 28.00 [13.50 to 34.00] | 144.00 [76.00 to 207.00] | 35.00 [1.00 to 69.00]
  CD8-TNF-α, Month 6: number analyzed (Participants) | 2 | 3 | 4
  CD8-TNF-α, Month 6 | 12.50 [1.00 to 24.00] | 1.00 [1.00 to 55.00] | 50.50 [16.50 to 86.50]
  CD8-TNF-α, Month 12: number analyzed (Participants) | 5 | 7 | 13
  CD8-TNF-α, Month 12 | 1.00 [1.00 to 23.00] | 28.00 [1.00 to 79.00] | 31.00 [1.00 to 69.00]
  CD8-TNF-α, Month 18: number analyzed (Participants) | 5 | 7 | 14
  CD8-TNF-α, Month 18 | 1.00 [1.00 to 1.00] | 60.00 [1.00 to 81.00] | 10.00 [1.00 to 219.00]
  CD8-TNF-α, Month 24: number analyzed (Participants) | 4 | 5 | 13
  CD8-TNF-α, Month 24 | 17.00 [1.00 to 42.00] | 78.00 [1.00 to 161.00] | 76.00 [21.00 to 142.00]
  CD8-TNF-α, Month 30: number analyzed (Participants) | 2 | 5 | 13
  CD8-TNF-α, Month 30 | 8.00 [1.00 to 15.00] | 1.00 [1.00 to 1.00] | 36.00 [1.00 to 82.00]
  CD8-TNF-α, Month 36: number analyzed (Participants) | 4 | 7 | 13
  CD8-TNF-α, Month 36 | 14.00 [1.00 to 38.50] | 1.00 [1.00 to 58.00] | 1.00 [1.00 to 21.00]
  CD8-TNF-α, Month 42 | 19.00 [1.00 to 23.00] | 1.00 [1.00 to 24.00] | 1.00 [1.00 to 27.00]
  CD8-TNF-α, Month 48: number analyzed (Participants) | 5 | 6 | 13
  CD8-TNF-α, Month 48 | 30.00 [1.00 to 59.00] | 1.00 [1.00 to 86.00] | 1.00 [1.00 to 30.00]
  CD8-TNF-α, Month 6/12/36 + 21 days: number analyzed (Participants) | 4 | 6 | 12
  CD8-TNF-α, Month 6/12/36 + 21 days | 26.00 [13.50 to 53.00] | 112.50 [81.00 to 194.00] | 46.00 [20.00 to 101.00]

30. Secondary Outcome: Frequency of Antigen-specific CD8 T-cells (Per 10E6) in Tests Identified as Producing at Least Two Out of Four Different Cytokines (for A/Vietnam/1194/2004 Strain)
Description: Among cytokines expressed after background reduction were cluster of differentiation 8 all doubles (CD8 all doubles), cluster of differentiation 40-ligand (CD40-L), interferon-gamma (IFN-γ), interleukin-2 (IL-2) and tumour necrosis factor-alpha (TNF-α). The flu strain assessed was H5N1 A/Vietnam/1194/2004.
Time Frame: At Months 6, 12, 18, 24, 30, 36, 42 and 48 and at Months 6/12/36 + 21 days
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: T-cells/million cells
Arm/Group | GSK1562902A M6 Group | GSK1562902A M12 Group | GSK1562902A M36 Group
Number analyzed (Participants) | 5 | 7 | 15
T-cells/million cells
  CD8-All doubles, Month 6: number analyzed (Participants) | 2 | 3 | 8
  CD8-All doubles, Month 6 | 33.00 [1.00 to 65.00] | 69.00 [1.00 to 91.00] | 1.00 [1.00 to 60.00]
  CD8-All doubles, Month 12: number analyzed (Participants) | 5 | 7 | 14
  CD8-All doubles, Month 12 | 26.00 [1.00 to 32.00] | 24.00 [21.00 to 106.00] | 24.00 [1.00 to 92.00]
  CD8-All doubles, Month 18 | 1.00 [1.00 to 1.00] | 63.00 [22.00 to 120.00] | 30.00 [1.00 to 87.00]
  CD8-All doubles, Month 24: number analyzed (Participants) | 4 | 5 | 13
  CD8-All doubles, Month 24 | 28.50 [7.50 to 50.00] | 33.00 [1.00 to 48.00] | 52.00 [1.00 to 256.00]
  CD8-All doubles, Month 30: number analyzed (Participants) | 2 | 5 | 13
  CD8-All doubles, Month 30 | 1.00 [1.00 to 1.00] | 46.00 [1.00 to 55.00] | 4.00 [1.00 to 85.00]
  CD8-All doubles, Month 36: number analyzed (Participants) | 4 | 7 | 13
  CD8-All doubles, Month 36 | 18.00 [1.00 to 183.00] | 96.00 [1.00 to 195.00] | 30.00 [1.00 to 71.00]
  CD8-All doubles, Month 42 | 1.00 [1.00 to 31.00] | 35.00 [1.00 to 38.00] | 26.00 [1.00 to 57.00]
  CD8-All doubles, Month 48: number analyzed (Participants) | 5 | 6 | 13
  CD8-All doubles, Month 48 | 12.00 [1.00 to 55.00] | 1.50 [1.00 to 20.00] | 19.00 [1.00 to 42.00]
  CD8-All doubles, Month 6/12/36 + 21 days: number analyzed (Participants) | 4 | 6 | 12
  CD8-All doubles, Month 6/12/36 + 21 days | 32.50 [14.00 to 47.00] | 133.50 [21.00 to 358.00] | 33.00 [1.00 to 210.50]
  CD8-CD40L, Month 6: number analyzed (Participants) | 2 | 3 | 8
  CD8-CD40L, Month 6 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 23.50]
  CD8-CD40L, Month 12: number analyzed (Participants) | 5 | 7 | 14
  CD8-CD40L, Month 12 | 12.00 [1.00 to 18.00] | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  CD8-CD40L, Month 18 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 12.00] | 1.00 [1.00 to 19.00]
  CD8-CD40L, Month 24: number analyzed (Participants) | 4 | 5 | 13
  CD8-CD40L, Month 24 | 21.50 [14.50 to 54.00] | 33.00 [8.00 to 48.00] | 17.00 [1.00 to 37.00]
  CD8-CD40L, Month 30: number analyzed (Participants) | 2 | 5 | 13
  CD8-CD40L, Month 30 | 1.00 [1.00 to 1.00] | 31.00 [1.00 to 49.00] | 1.00 [1.00 to 1.00]
  CD8-CD40L, Month 36: number analyzed (Participants) | 4 | 7 | 13
  CD8-CD40L, Month 36 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 18.00] | 4.00 [1.00 to 33.00]
  CD8-CD40L, Month 42 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 18.00] | 1.00 [1.00 to 20.00]
  CD8-CD40L, Month 48: number analyzed (Participants) | 5 | 6 | 13
  CD8-CD40L, Month 48 | 1.00 [1.00 to 28.00] | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  CD8-CD40L, Month 6/12/36 + 21 days: number analyzed (Participants) | 4 | 6 | 12
  CD8-CD40L, Month 6/12/36 + 21 days | 10.00 [1.00 to 37.50] | 1.00 [1.00 to 64.00] | 1.00 [1.00 to 28.50]
  CD8-IFN-γ, Month 6: number analyzed (Participants) | 2 | 3 | 8
  CD8-IFN-γ, Month 6 | 33.00 [1.00 to 65.00] | 22.00 [1.00 to 64.00] | 1.00 [1.00 to 32.00]
  CD8-IFN-γ, Month 12: number analyzed (Participants) | 5 | 7 | 14
  CD8-IFN-γ, Month 12 | 18.00 [1.00 to 26.00] | 67.00 [20.00 to 156.00] | 30.50 [1.00 to 93.00]
  CD8-IFN-γ, Month 18 | 1.00 [1.00 to 1.00] | 30.00 [1.00 to 149.00] | 2.00 [1.00 to 71.00]
  CD8-IFN-γ, Month 24: number analyzed (Participants) | 4 | 5 | 13
  CD8-IFN-γ, Month 24 | 10.00 [1.00 to 48.50] | 33.00 [16.00 to 79.00] | 51.00 [1.00 to 273.00]
  CD8-IFN-γ, Month 30: number analyzed (Participants) | 2 | 5 | 13
  CD8-IFN-γ, Month 30 | 1.00 [1.00 to 1.00] | 46.00 [1.00 to 55.00] | 1.00 [1.00 to 85.00]
  CD8-IFN-γ, Month 36: number analyzed (Participants) | 4 | 7 | 13
  CD8-IFN-γ, Month 36 | 23.00 [1.00 to 188.00] | 96.00 [24.00 to 159.00] | 4.00 [1.00 to 39.00]
  CD8-IFN-γ, Month 42 | 1.00 [1.00 to 23.00] | 35.00 [1.00 to 38.00] | 20.00 [1.00 to 41.00]
  CD8-IFN-γ, Month 48: number analyzed (Participants) | 5 | 6 | 13
  CD8-IFN-γ, Month 48 | 1.00 [1.00 to 12.00] | 1.00 [1.00 to 20.00] | 35.00 [1.00 to 49.00]
  CD8-IFN-γ, Month 6/12/36 + 21 days: number analyzed (Participants) | 5 | 6 | 12
  CD8-IFN-γ, Month 6/12/36 + 21 days | 27.50 [14.00 to 33.50] | 81.00 [21.00 to 293.00] | 25.50 [1.00 to 146.00]
  CD8-IL-2, Month 6: number analyzed (Participants) | 2 | 3 | 8
  CD8-IL-2, Month 6 | 3.50 [1.00 to 6.00] | 67.00 [1.00 to 68.00] | 28.00 [2.00 to 56.50]
  CD8-IL-2, Month 12: number analyzed (Participants) | 5 | 7 | 14
  CD8-IL-2, Month 12 | 25.00 [19.00 to 32.00] | 53.00 [8.00 to 79.00] | 7.50 [1.00 to 57.00]
  CD8-IL-2, Month 18 | 1.00 [1.00 to 1.00] | 47.00 [1.00 to 60.00] | 2.00 [1.00 to 45.00]
  CD8-IL-2, Month 24: number analyzed (Participants) | 4 | 5 | 13
  CD8-IL-2, Month 24 | 1.00 [1.00 to 19.50] | 12.00 [1.00 to 39.00] | 51.00 [1.00 to 114.00]
  CD8-IL-2, Month 30: number analyzed (Participants) | 2 | 5 | 13
  CD8-IL-2, Month 30 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 24.00] | 19.00 [1.00 to 113.00]
  CD8-IL-2, Month 36: number analyzed (Participants) | 4 | 7 | 13
  CD8-IL-2, Month 36 | 1.00 [1.00 to 138.50] | 64.00 [1.00 to 124.00] | 1.00 [1.00 to 33.00]
  CD8-IL-2, Month 42 | 1.00 [1.00 to 11.00] | 1.00 [1.00 to 38.00] | 20.00 [1.00 to 44.00]
  CD8-IL-2, Month 48: number analyzed (Participants) | 5 | 6 | 13
  CD8-IL-2, Month 48 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 22.00] | 1.00 [1.00 to 3.00]
  CD8-IL-2, Month 6/12/36 + 21 days: number analyzed (Participants) | 4 | 6 | 12
  CD8-IL-2, Month 6/12/36 + 21 days | 23.00 [15.50 to 30.00] | 103.50 [1.00 to 227.00] | 39.00 [1.00 to 104.00]
  CD8-TNF-α, Month 6: number analyzed (Participants) | 2 | 3 | 8
  CD8-TNF-α, Month 6 | 29.00 [1.00 to 57.00] | 25.00 [1.00 to 91.00] | 32.50 [1.00 to 46.00]
  CD8-TNF-α, Month 12: number analyzed (Participants) | 5 | 7 | 14
  CD8-TNF-α, Month 12 | 1.00 [1.00 to 1.00] | 24.00 [8.00 to 80.00] | 39.50 [1.00 to 69.00]
  CD8-TNF-α, Month 18 | 1.00 [1.00 to 1.00] | 63.00 [15.00 to 95.00] | 19.00 [1.00 to 71.00]
  CD8-TNF-α, Month 24: number analyzed (Participants) | 4 | 5 | 13
  CD8-TNF-α, Month 24 | 45.50 [26.50 to 61.00] | 37.00 [33.00 to 52.00] | 77.00 [1.00 to 200.00]
  CD8-TNF-α, Month 30: number analyzed (Participants) | 2 | 5 | 13
  CD8-TNF-α, Month 30 | 10.50 [1.00 to 20.00] | 1.00 [1.00 to 55.00] | 39.00 [2.00 to 85.00]
  CD8-TNF-α, Month 36: number analyzed (Participants) | 4 | 7 | 13
  CD8-TNF-α, Month 36 | 23.00 [1.00 to 133.00] | 111.00 [1.00 to 142.00] | 1.00 [1.00 to 67.00]
  CD8-TNF-α, Month 42 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 18.00] | 20.00 [1.00 to 57.00]
  CD8-TNF-α, Month 48: number analyzed (Participants) | 5 | 6 | 13
  CD8-TNF-α, Month 48 | 1.00 [1.00 to 12.00] | 1.00 [1.00 to 20.00] | 20.00 [1.00 to 29.00]
  CD8-TNF-α, Month 6/12/36 + 21 days: number analyzed (Participants) | 4 | 6 | 12
  CD8-TNF-α, Month 6/12/36 + 21 days | 15.50 [7.00 to 23.00] | 127.00 [21.00 to 227.00] | 7.50 [1.00 to 162.50]

31. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination. Grade 3 AE = an AE which prevented normal, everyday activities. Related = AE assessed by the investigator as related to the vaccination.
Time Frame: During the 30-day (Days 0-29) follow-up period after vaccination
Population: as for outcome 26
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A M12 Group | GSK1562902A M36 Group
Number analyzed (Participants) | 188 | 390
Participants
  Any AE(s) | 44 | 85
  Grade 3 AE(s) | 6 | 9
  Related AE(s) | 22 | 34

32. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: During the entire study period (From Month 12 up to Month 48)
Population: as for outcome 26
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A M6 Group | GSK1562902A M12 Group | GSK1562902A M36 Group
Number analyzed (Participants) | 219 | 188 | 437
Participants
  Month 12 to Month 48 | 14 | 13 | 28
  Month 42 to Month 48 | 2 | 3 | 4

ADVERSE EVENTS:
Time Frame: SAEs, AESIs : During the entire study period (From Month 12 to Month 48); Solicited local AEs: During the 7-day (Days 0-6) post-vaccination period for subjects boosted at Month 12 and Month 36; Solicited general AEs: During the 7-day (Days 0-6) post-vaccination period for subjects boosted at Month 12 and 36; Unsolicited AEs: During the 30-day (Days 0-29) follow-up period after vaccination.
Description: Non serious AEs (solicited local/ general/ unsolicited) were collected for M6 subset and are reported in study 109630 (NC T00449670) during which they received their booster vaccination.
Arm/Group | GSK1562902A M6 Group | GSK1562902A M12 Group | GSK1562902A M36 Group
All-Cause Mortality (participants affected / at risk) | 0/219 | 0/188 | 0/437
Serious Adverse Events (participants affected / at risk) | 14/219 | 13/188 | 28/437
Other Adverse Events (participants affected / at risk) | 0/0 | 169/188 | 336/437
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GSK1562902A M6 Group (N=219) | GSK1562902A M12 Group (N=188) | GSK1562902A M36 Group (N=437)
Appendicitis (Infections and infestations) | 1 | 1 | 3
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 1 | 3
Meniscus lesion (Injury, poisoning and procedural complications) | 0 | 0 | 4
Joint injury (Injury, poisoning and procedural complications) | 1 | 0 | 2
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 1
Chest pain (Hepatobiliary disorders) | 0 | 1 | 1
Cholecystitis chronic (Hepatobiliary disorders) | 1 | 1 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 2
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Appendicitis perforated (Infections and infestations) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Bipolar disorder (Psychiatric disorders) | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0
Choroidal detachment (Eye disorders) | 0 | 0 | 1
Chronic sinusitis (Infections and infestations) | 0 | 0 | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1
Dengue fever (Infections and infestations) | 1 | 0 | 0
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0
Endometriosis (Reproductive system and breast disorders) | 0 | 0 | 1
Excoriation (Injury, poisoning and procedural complications) | 0 | 1 | 0
Exostosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1
Intervertebral disc displacement (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 1
Morton's neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0
Normal tension glaucoma (Eye disorders) | 1 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 1
Optic neuritis (Nervous system disorders) | 0 | 0 | 1
Pericardial effusion (Cardiac disorders) | 1 | 0 | 0
Peritoneal adhesions (Gastrointestinal disorders) | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1
Pyelonephritis acute (Infections and infestations) | 0 | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Renal colic (Renal and urinary disorders) | 1 | 0 | 0
Renal cyst (Renal and urinary disorders) | 1 | 0 | 0
Retinal detachment (Eye disorders) | 0 | 0 | 1
Rhinitis (Infections and infestations) | 0 | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Salpingo-oophoritis (Infections and infestations) | 0 | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Viith nerve paralysis (Nervous system disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK1562902A M6 Group (N=0) | GSK1562902A M12 Group (N=188) | GSK1562902A M36 Group (N=437)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 48 (48) | 99 (100)
Chills (General disorders) | 0 | 26 (26) | 51 (51)
Erythema (Skin and subcutaneous tissue disorders) | 0 | 13 (13) | 28 (28)
Fatigue (General disorders) | 0 | 113 (113) | 216 (216)
Headache (Nervous system disorders) | 0 | 76 (77) | 139 (140)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 22 (22) | 54 (54)
Induration (General disorders) | 0 | 17 (17) | 23 (23)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 123 (123) | 235 (235)
Pain (General disorders) | 0 | 158 (158) | 306 (308)
Pyrexia (General disorders) | 0 | 17 (18) | 24 (24)
Swelling (General disorders) | 0 | 23 (23) | 44 (44)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.